CLINICAL TRIAL: NCT01589393
Title: OPtimal Timing of Thromboprophylaxis in Traumatic IntraCranial Haemorrhage (OPTTTICH Feasibility Study)
Acronym: OPTTTICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIHR-2009
Record Dates: First submitted 2012-04-26; First posted 2012-05-02 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2012-04

CONDITIONS: Traumatic Intracranial Haemorrhage
Keywords: Trauma; Thromboprophylaxis; Intracranial haemorrhage; Deep vein Thrombosis
MeSH Terms: conditions — Intracranial Hemorrhage, Traumatic; Wounds and Injuries; Intracranial Hemorrhages; Venous Thrombosis | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early initiation of thromboprophylaxis (Active Comparator): Early initiation of thromboprophylaxis with Enoxaparin between 36-48 hours post injury to day 5, followed by standard of care (DVT prophylaxis with Enoxaparin) starting day 6 post injury.
  Interventions: Drug: Enoxaparin
- Late initiation of thromboprophylaxis (Placebo Comparator): Initiation of placebo 36-48 hours post traumatic injury until day 5, then standard of care (DVT prophylaxis with Enoxaparin) starting on Day 6.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Enoxaparin — Enoxaparin 30 mg subcutaneously twice daily for six doses starting 36-48 hours post traumatic injury.
  Other Names: Lovenox
  Arms: Early initiation of thromboprophylaxis
Other: Placebo — 0.9% normal saline in equal volume to active comparator given subcutaneously twice daily starting 36-48 hours post traumatic injury for six doses.
  Arms: Late initiation of thromboprophylaxis

SUMMARY:
Victims of trauma with severe head injury who have bled into their brains are at high risk of developing blood clots in their legs. These blood clots can break off and travel through the bloodstream to the lungs causing death. Blood thinners can be given to patients to prevent blood clots from developing but this can leave patients at risk for additional bleeding in the brain causing further damage or death. The earlier blood thinners are started the more effective they are at preventing blood clots but some patients with severe head injury who have bled into their brains will develop further bleeding even if they do not receive blood thinners. Even though a growing body of research has shown that the majority of bleeding in the brain stops within the first 24 hours after injury and that it is safe to start blood thinners as early as 24 hours after injury, doctors are still waiting longer than 4 days to start blood thinners in these patients over concerns of worsening bleeding. In Canada, almost half of the patients with severe head injury do not receive blood thinners until at least five days after injury. Delays in starting blood thinners appear to put patients at increased risk of developing blood clots, unnecessarily. This study will compare the benefits of starting low-molecular weight heparin (LMWH), a type of blood thinner, early (less than 48 hours) versus the current practice (waiting until the 5th day after being injured) in preventing blood clots in patients who have bled into their brains after severe head injury. The investigators believe that starting LMWH earlier will be more effective in preventing blood clots without worsening any bleeding when compared to waiting to start blood thinners. This study is called OPTTTICH (Optimal Timing of Thromboprophylaxis in Traumatic IntraCranial Haemorrhage) and will be the largest Canadian investigator-initiated randomized control trial on blood clot prevention in trauma patients with severe head injury who have bled into their brains.

ELIGIBILITY:
Inclusion Criteria:

1. Multi-system trauma patients referred to the trauma service with a non-progressing tICH documented on 24-hour repeat head CT scan

Exclusion Criteria:

1. Less than 16 years of age
2. Unexpected to survive or to remain in hospital >72 hours
3. Known malignancy under active care at time of admission
4. Known DVT, PE, or other condition requiring anticoagulation at time of admission
5. Coagulopathy (defined as international normalized ratio (INR) values >1.5 times the upper limit of normal, or partial thromboplastin time (PTT) values >1.5 times the upper limit of normal) at 24 hours after admission
6. Platelet count <75 x 109/L at 24 hours after admission
7. Bilateral lower limb amputation
8. History of allergy to heparin or suspected or proven HIT
9. Limitation of life support or palliative care
10. Prior enrolment in this trial or currently in a confounding randomized trial
11. Pregnancy
12. Study drug (LMWH or placebo) not administered within 36-48 hours post-injury
13. Grade V liver or splenic injuries that have not received definitive care (e.g. embolization, surgical intervention) within 36-48 hours after injury
14. Persistent intracranial pressure >20 mm Hg
15. Spinal subdural haematoma or spinal epidural haematoma
16. Intracranial haemorrhage progression on 24-hour repeat CT head scan

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Proximal lower limb deep vein thrombosis (DVT) diagnosed by bilateral lower extremity compression ultrasound. | Maximum of 60 days or until hospital discharge.
  Ultrasounds will be performed within 72 hours of enrollment as well as twice weekly when in ICU and weekly thereafter. Non-compressibility of 1 or more proximal deep venous segments on compression US will be considered diagnostic. Each segment will be assessed as fully compressible, partially compressible, not compressible, or not well visualized. All positive ultrasounds will be recorded and stratified into above knee (proximal DVT) or below knee (distal DVT). Patients who have both proximal and distal vein thrombus will be classified as having proximal DVT.

SECONDARY OUTCOMES:
Non-intracranial bleeding | Maximum of 60 days or until hospital discharge.
  Non-intracranial bleeding events will be recorded and classified as either major or minor bleeding, according to a modified bleeding assessment tool adapted to our patient population.
Pulmonary Embolism | Maximum of 60 days or until hospital discharge
  Patients who develop clinical suspsicion of PE will have a helical CT chest. Pulmonary embolism will be diagnosed by the presence of an intraluminal filling defect detected in either the main,lobar,or segmental branches of the pulmonary artery. Patients with a high probability of PE on clinical grounds but with negative CT chest will undergo a ventilation-perfusion scan.
Intracranial haemorrhage progression (IHP). | Maximum of 60 days or until hospital discharge.
  If a Patient develops clinical evidence of neurological deterioration an emergent head CT scan will be performed.The CT scan will be reviewed by the blinded attending neuroradiologist. A comparison to the previous CT scan will be made and assessed for evidence of IHP. Intracranial haemorrhage progression will be defined as either 1) the development of a new haematoma, 2) any enlargement of an existing haematoma by an attending neuroradiologist's CT report, or 3) any progression of haematoma by the Marshall Head CT Classification System.

CONTACTS AND LOCATIONS:
Overall Officials: Niv Sne, MD FRCSC, Principal Investigator — Hamiltn Health Sciences/McMaster University
Locations (1):
- Hamilton Health Sciences- General site, Hamilton, Ontario, Canada